CLINICAL TRIAL: NCT01017731
Title: A Study to Evaluate the Relationship Between Ramucirumab (IMC-1121B) Therapy and Corrected QT (QTc) Interval Changes in Patients With Advanced Cancer
Brief Title: Study of Ramucirumab (IMC-1121B) Therapy and Corrected QT (QTc) Interval Changes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13915; CP12-0712 (Other: ImClone Systems); I4T-IE-JVBK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Cancer; Solid Tumor
Keywords: Advanced Solid tumor; Antibodies, Monoclonal; QTc; Metastatic; Malignant
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Ramucirumab; Moxifloxacin; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-1121B (Experimental): Active-control participants (first 16 participants) will receive one dose of moxifloxacin orally 7 days before the first treatment with ramucirumab. All participants will undergo triplicate electrocardiogram (ECG) tests (consisting of three individual ECGs performed consecutively within a period of 4 minutes) and vital signs at various times over the trial period.
  For Cycle 1, all participants will also receive 2 infusions of diphenhydramine before ramucirumab therapy (the first infusion is 1 day before therapy and the second infusion is 15 minutes before therapy). For Cycles 2, 3, and 4, all participants will receive diphenhydramine 15 minutes before ramucirumab therapy. For Cycle 5 and beyond, diphenhydramine infusions before ramucirumab therapy are at the investigator's discretion. Ramucirumab [10 milligrams per kilogram (mg/kg)] intravenously over 60 minutes, once every 3 weeks for minimum of 9 weeks without a break in between.
  Interventions: Biological: IMC-1121B; Drug: Moxifloxacin; Drug: Diphenhydramine

INTERVENTIONS:
Biological: IMC-1121B — IMC-1121B (Ramucirumab) 10 mg/kg intravenously (IV) over 60 minutes, once every 3 weeks for minimum of 9 weeks.
  Other Names: Ramucirumab; LY3009806
Drug: Moxifloxacin — Administered orally
Drug: Diphenhydramine — Administered IV

SUMMARY:
The purpose of this study is to determine if Ramucirumab (IMC-1121B) causes prolongation of the QT/QTc interval in participants with advanced cancer.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine if treatment with ramucirumab causes prolongation of the QTc/QT interval in participants with advanced cancer, to assess the safety and tolerability of ramucirumab therapy, and to evaluate the pharmacokinetic (PK) characteristics of ramucirumab

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically documented advanced or metastatic malignant cancer of solid tumor origin which has not responded to standard therapy or for which no standard therapy is available
* The participant has resolution of adverse events from prior anticancer therapies
* Performance status of 0 to 2
* The participant is ≥ 18 years of age
* The participant is able to provide informed written consent and is amenable to compliance with protocol schedules and testing
* The participant has adequate liver, kidney, blood, and blood clotting functions as defined in trial entrance criteria
* The participant agrees to use adequate contraception during the study period and for 8 weeks after the last dose of study treatment

Exclusion Criteria:

* The participant had anticancer therapy within 14 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* The participant had therapeutic radiotherapy within 14 days prior to entering the study
* The participant has ongoing side effects ≥ Grade 2 due to prior anticancer therapy
* The participant has brain or leptomeningeal metastases
* The participant has a history of uncontrolled or severe cardiac disease
* The participant has a history of severe congestive heart failure (CHF)
* The participant has a known history of arterial thrombotic events
* The participant has a known history of significant peripheral arterial disease (PAD)
* The participant has an implantable pacemaker or automatic implantable cardioverter defibrillator (AICD)
* The participant has a history of risk factors for ventricular tachycardia or Torsades de pointes (TdP) [for example, family history (parents or siblings) of long QT syndrome], history of fainting, unexplained loss of consciousness, or convulsions
* The participant has a systolic blood pressure (SBP) of > 150 millimeters of mercury (mmHg) or < 90 mmHg or a diastolic blood pressure (DBP) of < 45 or > 95 mmHg. (Participants with a history of hypertension who are receiving antihypertensive therapy are permitted on study provided blood pressure is within the parameters detailed above)
* The participant has a heart rate < 50 beats per minute (bpm) or > 100 bpm at rest
* The participant has a clinically relevant abnormality on the ECG, preventing an accurate measurement of the QT interval
* The participant is using a medication that is known to prolong the ECG QT interval
* The participant has a known allergy to any of the treatment components including fluoroquinolone antibiotics
* The participant has received an investigational new drug or device within 14 days prior to enrollment into this study (excluding placement of an intravenous access device)
* The participant has undergone major surgery within 28 days prior to enrollment
* The participant has known human immunodeficiency virus (HIV) infection
* The participant, if female, is pregnant or lactating
* The participant is receiving chronic daily treatment with aspirin [> 325 milligrams per day (mg/day)]
* The participant has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer, other noninvasive carcinoma, or in situ neoplasm
* The participant has psychological, familial, sociological, or geographical conditions which do not permit adequate study follow-up, compliance with the protocol, or signature of Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Providence, Rhode Island
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Olszanski AJ, Smith DC, Camacho LH, Thompson J, Ramalingam SS, Harvey RD, Campos L, Ferry D, Tang S, Gao L, Safran H. Electrocardiographic Characterization of Ramucirumab on the Corrected QT Interval in a Phase II Study of Patients With Advanced Solid Tumors. Oncologist. 2016 Apr;21(4):402-3. doi: 10.1634/theoncologist.2015-0467. Epub 2016 Mar 16. PMID 26984445

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 participants signed the informed consent.
Groups:
- IMC-1121B (Ramucirumab): Ramucirumab: 10 milligrams/kilogram (mg/kg) infused intravenously, every 3 weeks (Day 1 of every 21-day cycle). Treatment continued for a minimum of 9 weeks without a break in between until there was evidence of disease progression or intolerable toxicity.
  Diphenhydramine: For Cycle 1 only, 25 to 50 milligrams (mg) diphenhydramine infused intravenously 1 day before ramucirumab therapy. For Cycles 1, 2, 3, and 4, 25 to 50 mg diphenhydramine infused intravenously 15 minutes before ramucirumab therapy. For Cycle 5 and beyond, premedication with diphenhydramine was at the discretion of the investigator. Each participant was administered the same dose of diphenhydramine at all time points.
  Moxifloxacin: The first 16 participants enrolled received a single dose of moxifloxacin (400 mg tablet orally by mouth) 1 week prior to being treated with ramucirumab.
Period: Overall Study
Arm/Group | IMC-1121B (Ramucirumab)
Started | 68
Received at Least 1 Dose of Study Drug | 66
Completed | 60
Not Completed | 8
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety population: Participants who received any quantity of ramucirumab, regardless of their eligibility for the study.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 66
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 40
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  White | 60
  Black | 5
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 66
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 4
  Non-Hispanic or Latino | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Cycle 3 in QT/Corrected QT (QTc) Interval Prolongation in Participants
Description: All electrocardiogram (ECG) tests were performed in triplicate prior to ramucirumab treatment. QT is the interval between the Q and T waves and QTc is the QT corrected for heart rate using Fridericia's formula: QTc = QT/RR^0.33 where RR is the interval between 2 R waves. Each participant's mean QT/QTc value was calculated for each ECG test during Cycle 3 and compared to his/her mean pretreatment QT/QTc value. The greatest change from baseline during Cycle 3 was reported. QTc prolongation is defined as a QTc exceeding 10 milliseconds (msec) with a lower 90% confidence interval (CI) exceeding 5 msec at any postdose time points per the International Conference on Harmonization (ICH) E14 guidelines for non-thorough QT studies (ICH 2005; ICH 2008). Least squares (LS) mean was calculated using a linear mixed model for repeated measures (MMRM) and adjusted for serum concentration.
Time Frame: Baseline, Cycle 3 (1 cycle=21 days)
Population: Participants who received a full study dose of ramucirumab in Cycle 3 and had at least 1 pretreatment ECG and postinfusion ECG at scheduled times as specified in the protocol.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (msec)
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 66
milliseconds (msec) | 3.9132 [1.2880 to 6.5385]
Statistical Analysis 1: Comparison: IMC-1121B (Ramucirumab); Test type: Superiority or Other; p = 0.0161, Mixed Models Analysis — The p-value for QTc interval prolongation compared to baseline

2. Secondary Outcome: Number of Participants With Drug-Related Adverse Events (AEs)
Description: Data presented are the number of participants who experienced treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), Grade 3 or higher TEAEs, or adverse events (AEs) leading to discontinuation of treatment that were considered to be related to ramucirumab. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to data cut off (approximately 105.6 weeks)
Population: Safety population: participants who received any quantity of ramucirumab, regardless of their eligibility for the study.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 66
participants
  Related TEAE | 42
  Related SAE | 11
  Related Grade 3 or higher TEAE | 14
  Related AE leading to discontinuation | 6

3. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 1
Description: Maximum observed concentration of IMC-1121B (ramucirumab) in serum during Cycle 1 (1 cycle=21 days).
Time Frame: Cycle 1 [2.25 hours (h), 3.25 h, 4.25 h, 72 h, 168 h, 336 h postdose]
Population: Participants who received a full dose of ramucirumab and have evaluable Cmax data during Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 61
micrograms per milliliter (mcg/mL) | 485 (43)

4. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 1, Day 4
Description: Cmax was summarized once per cycle because participants only received 1 dose of IMC-1121B (ramucirumab) per cycle. Refer to secondary outcome measure 3 for Cmax during Cycle 1.
Time Frame: Approximately Week 1 (Cycle 1, Day 4)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 1, Day 8
Description: as for outcome 4
Time Frame: Approximately Week 2 (Cycle 1, Day 8)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 1, Day 15
Description: as for outcome 4
Time Frame: Approximately Week 3 (Cycle 1, Day 15)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 2
Description: Cmax was not calculated due to the sparse pharmacokinetic sampling employed on Cycle 2, Day 1.
Time Frame: Cycle 2 (predose and 1.25 hours postdose)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

8. Secondary Outcome: Maximum Concentration (Cmax) During Cycle 3
Description: The maximum observed serum concentration of IMC-1121B (ramucirumab) at steady state (Cmax,ss) during Cycle 3 (1 cycle=21 days).
Time Frame: Cycle 3 [predose and 1.25 hours (h), 2.25 h, 3.25 h, 4.25 h, 72 h, 168 h, 336 h, and 504 h postdose]
Population: Participants who received a full dose of ramucirumab and have evaluable Cmax data during Cycle 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 45
micrograms per milliliter (mcg/mL) | 571 (41)

9. Secondary Outcome: Area Under Concentration (AUC) During Cycle 1
Description: The area under the concentration versus time curve from time 0 to infinity [AUC(0-inf)] is reported during Cycle 1 (1 cycle=21 days).
Time Frame: Cycle 1 [2.25 hours (h), 3.25 h, 4.25 h, 72 h, 168 h, 336 h postdose]
Population: Participants who received a full dose of ramucirumab and have evaluable AUC data during Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliter (h*mcg/mL)
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 58
hours*micrograms/milliliter (h*mcg/mL) | 67400 (38)

10. Secondary Outcome: Area Under Concentration (AUC) During Cycle 1, Day 4
Description: AUC was summarized once per cycle because participants only received 1 dose of IMC-1121B (ramucirumab) per cycle. Refer to secondary outcome measure 9 for AUC during Cycle 1 (Day 1 through Day 15).
Time Frame: Approximately Week 1 (Cycle 1, Day 4)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

11. Secondary Outcome: Area Under Concentration (AUC) During Cycle 1, Day 8
Description: as for outcome 10
Time Frame: Approximately Week 2 (Cycle 1, Day 8)
Population: No participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

12. Secondary Outcome: Area Under Concentration (AUC) During Cycle 1, Day 15
Description: as for outcome 10
Time Frame: Approximately Week 3 (Cycle 1, Day 15)
Population: No participants analyzed.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

13. Secondary Outcome: Area Under Concentration (AUC) During Cycle 2, Day 1
Description: AUC was not calculated due to the sparse pharmacokinetic sampling employed on Cycle 2, Day 1.
Time Frame: Approximately Week 1 (Cycle 2, Day 1)
Population: No participants were analyzed.
Groups:
- IMC-1121B (Ramucirumab): Ramucirumab: 10 milligrams/kilogram (mg/kg) infused intravenously over 1 hour, every 3 weeks (Day 1 of every 21-day cycle). Treatment continued for a minimum of 9 weeks without a break in between until there was evidence of disease progression or intolerable toxicity.
  Diphenhydramine: 25 to 50 milligrams (mg) administered intravenously 1 day before each administration of ramucirumab for Cycles 1 to 4. For Cycle 5 and beyond, premedication with diphenhydramine was at the discretion of the investigator. Each participant was administered the same dose of diphenhydramine at all time points.
  Moxifloxacin: The first 16 participants enrolled received a single dose of moxifloxacin (400 mg tablet orally by mouth) 1 week prior to being treated with ramucirumab.
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0

14. Secondary Outcome: Area Under Concentration (AUC) During Cycle 3
Description: The area under the concentration versus time curve over the dosing interval at steady state [AUC(tau,ss)] is reported during Cycle 3 (1 cycle=21 days).
Time Frame: Cycle 3 [predose and 1.25 hours (h), 2.25 h, 3.25 h, 4.25 h, 72 h, 168 h, 336 h, and 504 h postdose]
Population: Participants who received a full dose of ramucirumab and have evaluable AUC data during Cycle 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliter (h*mcg/mL)
Arm/Group | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 38
hours*micrograms/milliliter (h*mcg/mL) | 69900 (41)

ADVERSE EVENTS:
Arm/Group | IMC-1121B (Ramucirumab)
Serious Adverse Events (participants affected / at risk) | 32/66
Other Adverse Events (participants affected / at risk) | 61/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) (N=66)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Disease progression (General disorders) | 6 (9)
Infusion related reaction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) (N=66)
Anaemia (Blood and lymphatic system disorders) | 4 (6)
Hypothyroidism (Endocrine disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 16 (18)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 16 (21)
Nausea (Gastrointestinal disorders) | 21 (36)
Vomiting (Gastrointestinal disorders) | 16 (22)
Asthenia (General disorders) | 7 (7)
Chills (General disorders) | 9 (9)
Fatigue (General disorders) | 21 (27)
Oedema peripheral (General disorders) | 11 (19)
Pyrexia (General disorders) | 10 (11)
Seasonal allergy (Immune system disorders) | 4 (4)
Blood creatinine increased (Investigations) | 4 (9)
Abnormal loss of weight (Metabolism and nutrition disorders) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 22 (24)
Dehydration (Metabolism and nutrition disorders) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (10)
Dizziness (Nervous system disorders) | 10 (12)
Headache (Nervous system disorders) | 20 (29)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.